CLINICAL TRIAL: NCT03079882
Title: VisR Ultrasound for Noninvasively Monitoring Renal Allograft Health
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-2934; 1R01DK107740 (NIH)
Record Dates: First submitted 2017-02-17; First posted 2017-03-15 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-05

CONDITIONS: Renal Transplant Failure
Keywords: Ultrasound; Viscoelasticity; Viscoelastic Response (VisR) Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Living Donor Recipients: Recipients of renal transplants with the transplanted organ originating from living donors
- Deceased Donor Recipients: Recipients of renal transplants with the transplanted organ originating from deceased donors

SUMMARY:
Ten percent of American adults, more than 20 million people, have chronic kidney disease, which in the advanced state of end stage renal disease is most desirably and cost-effectively treated by kidney transplantation. However, 20-30% of transplanted kidneys fail in living recipients by 10 years, owing largely to insufficient monitoring methods. The goal of the proposed research is to improve noninvasive kidney transplant monitoring using a new ultrasound-based imaging method called Viscoelastic Response (VisR) ultrasound.

DETAILED DESCRIPTION:
Renal transplantation is the most desirable and cost effective treatment for end stage renal disease, but 20-30% of allografts fail in living recipients by 10 years, and prolonging graft health is one of the major unmet needs for transplant patients. Although graft health is extended by preemptive treatments that prevent irreversible damage, intervention is inadequately motivated by current transplant monitoring methods. Noninvasive methods, including changes in serial serum creatinine levels, lack sensitivity and specificity. In the absence of reliable noninvasive biomarkers, invasive biopsy remains the standard for assessing transplant health, but surveillance or "protocol" biopsies are associated with morbidity and cost and are therefore controversial in stable, unsensitized patients. The lack of a demonstrated, noninvasive biomarker for allograft health - one that identifies early graft degeneration with sufficient sensitivity and specificity to motivate appropriate biopsy and enable timely intervention - represents a major gap in renal transplant management.

To fill this gap, the proposed re-search aims to demonstrate Viscoelastic Response (VisR) ultrasound, a novel acoustic radiation force (ARF)-based technology that noninvasively interrogates the viscoelastic properties of tissue, for monitoring renal allograft health. The investigators hypothesize that in vivo VisR ultrasound delineates renal allograft dysfunction earlier and with greater sensitivity and specificity than serum creatinine concentration in renal allograft recipients.

To test this hypothesis, the investigators will determine which VisR outcome metrics detect renal allograft dysfunction clinically by performing serial VisR imaging in living donor (LD) and deceased donor (DD) transplant recipients. Imaging results will be compared to biopsy findings to determine VisR's ability to detect dysfunction. The investigators will also compare serial VisR and serum creatinine outcomes in terms of ability to detect renal allograft dysfunction and the timeliness of detection.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Selected by treating physician to be in need of renal transplant surgery
3. Ability to provide informed consent
4. Ability to communicate with pertinent staff
5. Ability to understand and comply with study requirements

Exclusion Criteria:

1. Inability to provide valid consent
2. Inability to communicate with pertinent staff
3. Inability to remain motionless for at least 20 minutes
4. Renal transplant deeper than 4 cm

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This unblinded, open-label, exploratory study will be conducted in 100 consecutively evaluable patients (50 with renal allografts from living donors and 50 with allografts from deceased donors). Patients will be recruited from those already undergoing renal transplant surgery for end stage renal disease based on the standard of care at UNC Hospitals. Potential study participants will be patients 18 years of age or older who have been selected by their treating physician to be in need of renal transplant surgery for end stage renal disease at University of North Carolina Hospitals' Nephrology Transplant clinic. Participants will be enrolled in two groups, as living or deceased donor recipients. There will be no intervention beyond VisR ultrasound imaging.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
VisR AUC value | at time of clinically indicated biopsy
  AUC for VisR to detect positive biopsy finding (indiscriminate of type)

SECONDARY OUTCOMES:
AUC for the ability of change in serum creatinine level to detect positive biopsy finding | at time of clinically indicated biopsy
  Receiver operating characteristic (ROC) curve analysis will be performed using pathology findings as the gold standard. From the ROC curve, AUC will be calculated.
AUC for the ability of change in VisR Tau value to detect positive biopsy finding | at time of clinically indicated biopsy
  Receiver operating characteristic (ROC) curve analysis will be performed using pathology findings as the gold standard. From the ROC curve, AUC will be calculated.
AUC for the ability of change in VisR Relative Elasticity value to detect positive biopsy finding | at time of clinically indicated biopsy
  Receiver operating characteristic (ROC) curve analysis will be performed using pathology findings as the gold standard. From the ROC curve, AUC will be calculated.
AUC for the ability of change in VisR Relative Viscosity value to detect positive biopsy finding | at time of clinically indicated biopsy
  Receiver operating characteristic (ROC) curve analysis will be performed using pathology findings as the gold standard. From the ROC curve, AUC will be calculated.
Change in serum creatinine level | 1-2 weeks, 4 weeks, 2 months, 3 months, 6 months, 9 months, 12 months, and then every 4 months after transplantation until time of clinically indicated biopsy or 3 years after transplantation, which ever comes first
  serum creatine will be measured serially, consistent with clinical indication, and change in level from time point to time point will be recorded.
Change in VisR Tau value | 1-2 weeks, 4 weeks, 2 months, 3 months, 6 months, 9 months, 12 months, and then every 4 months after transplantation until time of clinically indicated biopsy or 3 years after transplantation, which ever comes first
  VisR Tau will be measured serially, and change in values from time point to time point will be recorded.
Change in VisR Relative Elasticity value | 1-2 weeks, 4 weeks, 2 months, 3 months, 6 months, 9 months, 12 months, and then every 4 months after transplantation until time of clinically indicated biopsy or 3 years after transplantation, which ever comes first
  VisR Relative Elasticity will be measured serially, and change in values from time point to time point will be recorded.
Change in VisR Relative Viscosity value | 1-2 weeks, 4 weeks, 2 months, 3 months, 6 months, 9 months, 12 months, and then every 4 months after transplantation until time of clinically indicated biopsy or 3 years after transplantation, which ever comes first
  VisR Relative Viscosity will be measured serially, and change in values from time point to time point will be recorded.
AUC for the ability of VisR-derived Tau to detect positive biopsy finding | at time of clinically indicated biopsy
  Tau represents the relaxation time constant for constant stress in a Voigt material and reflects the ratio of viscous to elastic properties of the kidney in the examined region.
AUC for the ability of VisR-derived Relative Elasticity to detect positive biopsy finding | at time of clinically indicated biopsy
  Relative elasticity qualitatively represents the tissue elastic modulus relative to the applied force amplitude
AUC for the ability of VisR-derived Relative Viscosity to detect positive biopsy finding | at time of clinically indicated biopsy
  Relative viscosity qualitatively represents the tissue viscous modulus relative to the applied force amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Caterina M Gallippi, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No